CLINICAL TRIAL: NCT03700203
Title: Cardiac Arrest Pursuit Trial With Unique Registration and Epidemiologic Surveillance
Acronym: CAPTURES
Status: Recruiting | Type: Observational
Sponsor: Seoul National University Hospital (Other)
Collaborators: Korean Center for Disease Control and Prevention (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2017NE330060
Record Dates: First submitted 2018-08-21; First posted 2018-10-09 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2025-12

CONDITIONS: Cardiac Arrest, Out-Of-Hospital
Keywords: Cardiac Arrest
MeSH Terms: conditions — Out-of-Hospital Cardiac Arrest; Heart Arrest

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Early cardiac arrest patients: Cases will be consecutive adult patients with EMS-treated OHCA and transport to the 14 emergency departments of participating hospitals. A prospective OHCA patient cohort will be developed and all survived OHCA cases will be followed at 1-month and 6-month after ED discharge by telephone. During the study period, the investigators aim to recruit a total 1,780 cases (200 cases between September 2017 and August 2018, 600 cases between September 2018 and August 2020, 80 cases between September 2020 and December 2020, and 900 cases between January 2021 and December 2023).
- Matched community-based controls: Matched community-based controls (2:1 matching) will be selected from two health screening centers. Controls are those who visit the participating health screening centers for their annual routine physical examinations. During the study period, the investigators aim to recruit a total 3,560 controls (400 controls between September 2017 and August 2018, 1200 controls between September 2018 and August 2020, 160 controls between September 2020 and December 2020, and 1800 controls between January 2021 and December 2023).

SUMMARY:
Identification of Causes and Risk Factors for Out-of-Hospital Cardiac Arrest through Development of Prediction Model and Novel Biomarkers

Study Objectives:

1. To identify causes and risk factors of OHCA incidence that are associated with chronic diseases and health behaviors
2. To identify high risk population for OHCA incidence through development of a prediction model
3. To develop novel biomarkers associated with OHCA incidence, survival, and disabilities

DETAILED DESCRIPTION:
Study design: Multicenter case-control study, 14 tertiary teaching hospital emergency departments in Korea

Study period: September 2017 to December 2023 (75 months)

Study population: Early cardiac arrest patients aged between 19 and 79 (1,780 cases) and their age-, gender-, and urban/rural area-matched community controls (3,560 cases).

* Cases will be consecutive adult patients with EMS-treated OHCA and transport to the 14 emergency departments of participating hospitals. A prospective OHCA patient cohort will be developed and all survived OHCA cases will be followed at 1-month, 6-month, and 12-month after ED discharge by telephone. During the study period, the investigators aim to recruit a total 1,780 cases (200 cases between September 2017 and August 2018, 600 cases between September 2018 and August 2020, 80 cases between September 2020 and December 2020, and 900 cases between January 2021 and December 2023).
* matched community-based controls (2:1 matching) will be selected from two health screening centers. Controls are those who visit the participating health screening centers for their annual routine physical examinations. During the study period, the investigators aim to recruit a total 3,560 controls (400 controls between September 2017 and August 2018, 1200 controls between September 2018 and August 2020, 160 controls between September 2020 and December 2020, and 1800 controls between January 2021 and December 2023).

Data collection: Following data will be collected for both cases and controls.

* Clinical data: Basic demographic and clinical outcomes will be retrieved from medical records.
* Survey data: Comorbidity, family history of selected diseases, lifestyle behaviors (including smoking, alcohol, physical activity, sleeping, nutrition, marital status, occupation), and history of selected chronic diseases data will be collected.
* Blood samples: The investigators aim to develop both clinical and behavioral (including nutrition, alcohol, and smoking) biomarkers of OHCA. The investigators also plan to further develop OHCA biomarkers using proteomics, genomics, and metabolomics.
* Follow-ups: All survived OHCA cases will be followed-up at 1-month, 6-month, and 12-month after ED discharge and their survival, disability, and quality of life outcomes will be collected by telephone.

ELIGIBILITY:
Inclusion Criteria:

* 19 to 79 years old
* Out-of-hospital-cardiac arrest providing resuscitation at the site and visiting the emergency department of the participating hospital or transporting from another hospital emergency room (EMS-treated OHCA)
* The cardiac arrest event must not have been predicted for 24 hours before the incident

Exclusion Criteria:

* People who do not consent to personal information and blood supply for research
* Trauma, submersion, poisoning, hanging, suffocation, or other causes of external causes directly contribute to the cardiac arrest
* Patients with a terminal condition known to have no further treatment plans due to malignancy, neurological disease, respiratory disease, rheumatic disease, hematologic disease, renal disease or infectious disease. The terminal condition had to be checked by a doctor or recorded in medical records.
* "Do not have a resuscitation" card or record issued by a doctor.
* Hospice setting at the time of acute cardiac arrest for terminal illness or other reasons.
* pregnant patient
* With a family cannot provide information about patient
* Without a family
* Patients who were transported after admission at the other hospital
* Foreign patients

Ages: 19 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: * Cases will be consecutive adult patients with EMS-treated OHCA and transport to the 14 emergency departments of participating hospitals.
  * Matched community-based controls (2:1 matching) will be selected from two health screening centers. Controls are those who visit the participating health screening centers for their health screening program.
Sampling Method: Probability Sample
Enrollment: 5340 (Estimated)
Dates: Start 2017-09-07 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of Participants With Out-of-hospital Cardiac Arrests | A total 1,780 cases (200 cases between September 2017 and August 2018, 600 cases between September 2018 and August 2020, 80 cases between September 2020 and December 2020, and 900 cases between January 2021 and December 2023)
  Number of participants with out-of-hospital cardiac arrests, from 19 to 79 years old.

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

REFERENCES:
- [Derived] Jung E, Ryu HH, Ro YS, Cha KC, Shin SD, Hwang SO. Interactions between Sleep Apnea and Coronary Artery Disease on the Incidence of Sudden Cardiac Arrest: A Multi-Center Case-Control Study. Yonsei Med J. 2023 Jan;64(1):48-53. doi: 10.3349/ymj.2022.0417. PMID 36579379